CLINICAL TRIAL: NCT01221259
Title: A Randomized, Double-blind, Placebo-controlled, Sequential Ascending, Single-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of E2212 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: E2212-A001-001
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug E2212 (Experimental)
  Interventions: Drug: E2212
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: E2212 — single ascending doses ranging from 10mg to 250mg
  Arms: Drug E2212
Drug: placebo — a single dose of matching placebo
  Arms: Placebo

SUMMARY:
This study is designed as a single ascending dose study in healthy subjects to evaluate safety, tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) in plasma and Cerebrospinal (CSF) following single oral doses of E2212.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women of non-child bearing potential age 18 and 55 years old at the time of Screening;
2. Body mass index (BMI) 18 and 30 kg/m2 at Screening;
3. Are willing and able to comply with all aspects of the protocol; and
4. Provide written informed consent.

Exclusion Criteria:

1. Clinically important abnormalities on physical examination, vital signs or clinical laboratories.
2. History of serious medical illness
3. Smoking or use of tobacco-containing products within past 3 months
4. History of alcohol or drug abuse within past 2 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single ascending oral doses of E2212 in healthy subjects. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Philip Lee, Md, Principal Investigator — Quintiles Phase One Service
Locations (1):
- Overland Park, Kansas, United States